CLINICAL TRIAL: NCT05839340
Title: Neurally Adjusted Ventilatory Assist for Neonates With Congenital Diaphragmatic Hernias
Acronym: NAN-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: St George's, University of London (Other)
Responsible Party: Principal Investigator, Anne Greenough, Professor of Neonatology and Clinical Respiratory Physiology, King's College Hospital NHS Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 319769
Record Dates: First submitted 2023-04-07; First posted 2023-05-03 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Intervention Model Description: Dual Centre Randomised Cross-Over Trial. Infants that meet inclusion criteria will be randomised to be ventilated with either NIV-NAVA or ACV for four hours, followed by the second mode of ventilation. There will be a 20-minute stabilisation period between ventilatory methods.
Masking Description: Due to practical limitations, the trial will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurally Adjusted Ventilatory Assist (Experimental): Infants will first be ventilated with NAVA for four hours. Following this, they will undergo a 20-minute stabilisation period prior to ventilating with assist control ventilation (ACV).
  Interventions: Device: Neurally Adjusted Ventilatory Assist; Device: Assist Control Ventilation
- Assist Control Ventilation (ACV) (Experimental): Infants will first be ventilated with ACV for four hours. Following this, they will undergo a 20-minute stabilisation period prior to ventilating with non-invasive neurally adjusted ventilatory assist.
  Interventions: Device: Neurally Adjusted Ventilatory Assist; Device: Assist Control Ventilation

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist — NAVA uses electrical signals of the diaphragm to deliver a proportional pressure of oxygen, to which proportion is set by the clinician as the NAVA level.
  Other Names: Assist Control Ventilation
Device: Assist Control Ventilation — ACV delivers fixed oxygen pressure set by the clinician at the start of each inspiratory breath.

SUMMARY:
Congenital Diaphragmatic Hernias (CDH) are typically repaired surgically in the first few days of a neonate's life. Following surgical repair, infants usually require ventilatory support to ensure adequate oxygenation. Traditionally assist control ventilation (ACV) has been used to support neonates with CDH. Due to delivering a fixed pressure of oxygen, ACV has been associated with barotrauma and long-term lung damage. A more recent approach to ventilation is non-invasive neurally adjusted ventilatory assist (NIV-NAVA). NIV-NAVA uses electrical signals of the diaphragm to deliver a proportional pressure of oxygen. Our dual-centre randomised cross-over trial aims to investigate the efficacy of NIV-NAVA compared to ACV for supporting neonates with CDH.

DETAILED DESCRIPTION:
Background:

Congenital Diaphragmatic Hernias (CDH) are typically repaired surgically in the first few days of a neonate's life. Following surgical repair, infants usually require ventilatory support to ensure adequate oxygenation. Traditionally assist control ventilation (ACV) has been used to support neonates with CDH. Due to delivering a fixed pressure of oxygen, ACV has been associated with barotrauma and long-term lung damage. A more recent approach to ventilation is non-invasive neurally adjusted ventilatory assist (NIV-NAVA). NIV-NAVA uses electrical signals of the diaphragm to deliver a proportional pressure of oxygen. Evidence suggests that NAVA may reduce physiological parameters associated with lung pressure and hence reduce the risk of iatrogenic lung injury.

Aims:

Our aim is to compare the oxygenation index (OI) of neonates with CDH, ventilated with ACV and NIV-NAVA. The OI is calculated as the fractured of inspired oxygen x mean airway pressure x partial pressure of oxygen/100. The oxygenation index is used as a marker of hypoxic respiratory failure in infants with CDH and forms the basis of the criteria to administer nitric oxide.

Methods:

Our investigation is a dual-centre randomised cross-over trial. Infants will be identified and parents counselled in the first few days following delivery. Neonates that meet inclusion criteria will be randomised to receive either NIV-NAVA or ACV first, followed by the other method of ventilation. Infants will be stabilised on ACV one-hour prior to entering the trial. On entry into the trial, they will receive 4-hours of each ventilatory method with a 20-minute stabilisation break in between.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with congenital diaphragmatic hernia more than 34-weeks gestation

Exclusion Criteria:

* Receiving Nitric Oxide
* Requiring an FIO2 more than 80% to maintain SpO2: 85-95%.
* Severe chromosomal abnormality
* Severe cardiac anomalies requiring corrective surgery
* Renal anomalies
* Skeletal deformities suspected to impede thoracic or lung development
* Severe central nervous system anomalies suspected to impede diaphragmatic signalling
* Use of neuromuscular blocking agents
* Contraindication to nasogastric tube insertion

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Oxygenation Index (OI) | Infants will receive each mode of ventilation for four hours. OI will be recorded every 5-minutes for the final 30-minutes of each ventilation period. The OI will be averaged over the 30-minute time frame. This average OI will then be compared.
  Oxygenation Index is calculated as MAP x FIO2 x PaO2/100. MAP is the mean airway pressure. FIO2 represents the concentration of inspired oxygen and PAO2 is the partial pressure of oxygen. The OI is a reliable indicator of lung function, previous research has shown its use in the prognostication of neonates with CDH.

SECONDARY OUTCOMES:
Respiratory Severity Score (RSS) | RSS will be recorded every 5-minutes for the final 30-minutes that the infant is on each ventilation mode. This will be compared to their baseline 30-minutes pre-randomisation and between ventilation modes.
  The respiratory severity score is calculated as RSS = FIO2 x MAP. Where FIO2 represents the fraction of inspired oxygen and MAP is the mean airway pressure. In one multivariate analysis of 59 infants with CDH, RSS was an effective prognostic marker.

OTHER OUTCOMES:
Mean Airway Pressure (MAP) | MAP will be recorded every 5-minutes for the final 30-minutes that the infant is on each ventilation mode. This will be compared to their baseline 30-minutes pre-randomisation and between ventilation modes.
  The MAP is mean pressure the lungs are exposed to during inspiration and expiration. Mean airway pressure is one of the main determinants of oxygenation.
Fraction of Inspired Oxygen (FIO2) | FIO2 will be recorded every 5-minutes for the final 30-minutes that the infant is on each ventilation mode. This will be compared to their baseline 30-minutes pre-randomisation and between ventilation modes.
  The FIO2 is the concentration of oxygen delivered expressed as a percentage.
Peak Inspiratory Pressure (PIP) | PIP will be recorded every 5-minutes for the final 30-minutes that the infant is on each ventilation mode. This will be compared to their baseline 30-minutes pre-randomisation and between ventilation modes.
  Peak Inspiratory Pressure is defined as the pressure reached at the end of inspiration.
Morphine Equivalent Use | The cumulative total of morphine used during the four-hour period on each ventilation mode will be calculated. This will be compared between ventilation modes.
  Analgesic medication will be used with a basal-bolus regimen with the option for as required analgesia based on perceived pain and agitation.
Midazolam Equivalent Use | The cumulative total of midazolam, or equivalent benzodiezapine, used during the four-hour period on each ventilation mode will be calculated. This will be compared between ventilation modes
  Cumulative midazolam use on each ventilatory method will be calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Kings College Hospital, London
  - St. George's University Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Requests for individual participant data will be reviewed by the principal investigator. On request, data will be made available to other researchers 6-months following trial cessation. Parents will be consented to share their child's data for research purposes. All data will be anonymised on entry into the trial so no individual data point will be recognisable.
Supporting Information: Study Protocol, ICF
Time Frame: It is our intent that the NAN-C protocol will be published, following SPIRIT guidelines, following the start of the trial.
  At present, there are no plans to grant public access to the full protocol, participant-level data set or statistical code. For 6-months following publication of the final study results, investigators will be granted priority for secondary data analyses. Following this period, requests for de-identified data will be considered. Requests for data presented in the final paper should be submitted via email to Professor Anne Greenough.
Access Criteria: Requests for data presented in the final paper should be submitted via email to Professor Anne Greenough.

REFERENCES:
- [Derived] Poole G, Harris C, Shetty S, Dassios T, Jenkinson A, Greenough A. Study protocol for a randomised cross-over trial of Neurally adjusted ventilatory Assist for Neonates with Congenital diaphragmatic hernias: the NAN-C study. Trials. 2024 Jan 20;25(1):72. doi: 10.1186/s13063-023-07874-0. PMID 38245741